CLINICAL TRIAL: NCT02791841
Title: The Effectiveness of Intervention for Developmental Dyslexia: The Rhythmic Reading Training Compared With Hemisphere-Specific Stimulation and Action Video Games
Brief Title: Comparison of Interventions for Developmental Dyslexia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: IRCCS Eugenio Medea (Other)
Responsible Party: Principal Investigator, Alice Cancer, PhD candidate, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRT-VHSS-AVG
Record Dates: First submitted 2016-05-26; First posted 2016-06-07 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Developmental Dyslexia
Keywords: Reading; Developmental Dyslexia,; Music; Rhythm; Action Video Games; Hemisphere-Specific Stimulation
MeSH Terms: conditions — Dyslexia

ARMS (3):
- RRT (Experimental): Rhythmic Reading Training, administered for 13 hours over 9 days (two 45-minute training sessions per day).
  Interventions: Behavioral: Rhythmic Reading Training
- VHSS+AVG (Experimental): Visual Hemispheric-Specific Stimulation + Action Video Games, administered for 13 hours over 9 days (two 45-minute training sessions per day).
  Interventions: Behavioral: Visual Hemispheric-Specific Stimulation + Action Video Games
- AVG (Experimental): Action Video Games only, administered for 13 hours over 9 days (two 45-minute training sessions per day).
  Interventions: Behavioral: Action Video Games

INTERVENTIONS:
Behavioral: Rhythmic Reading Training — RRT is a child-friendly computerized reading training program designed for Italian students with DD aged 8-14 yrs. The main feature of this intervention is the integration of a traditional remediation approach (sublexical treatment) with rhythm processing. Therefore, all reading exercises are characterized by a rhythmic accompaniment with gradually increasing speed.
  Other Names: RRT
  Arms: RRT
Behavioral: Visual Hemispheric-Specific Stimulation + Action Video Games — This training combines Visual Hemisphere-Specific Stimulation (VHSS) according to Bakker's Balance Model, and Action Video-Games (AVG). Hemispheric-specific stimulation is carried out by tachistoscopic presentation of words to a visual hemifield in order to selectively stimulate right-hemisphere perceptual analysis or left-hemisphere linguistic anticipation. A computerized program is used, in which the word is flashed and presented for less than 350 ms only if the child clicks on the mouse at the exact moment a dot is crossing a central target (control of eye position and fixation).
  AVG training involves dyslexic participants in a video-game training, specifically aimed at improving visuo-spatial attentional abilities. A commercial WiiTM video game from UbisoftTM (suitable for children age 7 and older by the Pan European Game Information) called 'Rayman Raving Rabbids' is used.
  Other Names: VHSS+AVG
  Arms: VHSS+AVG
Behavioral: Action Video Games — AVG training involves dyslexic participants in a video-game training, specifically aimed at improving visuo-spatial attentional abilities. A commercial WiiTM video game from UbisoftTM (suitable for children age 7 and older by the Pan European Game Information) called 'Rayman Raving Rabbids' is used.
  Other Names: AVG
  Arms: AVG

SUMMARY:
The purpose of the present study is to compare the effectiveness of Rhythmic Reading Training (RRT), a computer-assisted intervention method that combines sublexical reading exercises with rhythm processing, and that of an intervention resulting from the combination of two yet validated treatments for DD, namely, Bakker's Visual Hemisphere-Specific Stimulation (VHSS) and the Action Video Game Training (AVG). Finally, the effectiveness of the administration of only AVG is intended to be compared to other treatments. All interventions are administered for 13 hours over 9 days to a group of Italian students with DD aged 8-12.

ELIGIBILITY:
Inclusion Criteria:

* having been diagnosed with DD (ICD-10 code: F81.0) on the basis of standard inclusion and exclusion criteria (ICD-10: World Health Organization, 1992) and of the diagnosis procedure followed in the Italian practice

Exclusion Criteria:

* presence of comorbidity with other neuropsychiatric or psychopathological conditions (whereas comorbidity with other learning disabilities were allowed)
* having been involved in previous reading intervention programs

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-06 (Actual); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Text reading | 3 weeks
  The ability to read aloud a text was assessed using the Italian standardized test 'New MT reading tests for junior high school' (Nuove prove di lettura MT per la scuola media inferiore), which provides accuracy and speed scores in reading aloud age-normed texts.
Word reading | 3 weeks
  The ability to read aloud lists of words was assessed using the following Italian standardized tests: 'Assessment battery for Developmental Dyslexia and Dysorthography-2' (Batteria per la valutazione della dislessia e disortografia evolutiva - DDE-2), in which speed and accuracy scores were computed for word reading (4 lists of 28 words each with different lengths and frequency of use); 'Word and pseudo-word reading test' (WPRT, Prova di lettura di parole e non parole), in which speed and accuracy scores were computed for word reading (4 lists of 30 words varying according to length: short vs. long and frequency of use: low vs. high frequency).
Pseudo-word reading | 3 weeks
  The ability to read aloud lists of pseudo-words was assessed using the following Italian standardized tests: 'Assessment battery for Developmental Dyslexia and Dysorthography-2' (Batteria per la valutazione della dislessia e disortografia evolutiva - DDE-2), in which speed and accuracy scores were computed for pseudo-word reading (2 lists of 16 pseudo-words each with different lengths); 'Word and pseudo-word reading test' (WPRT, Prova di lettura di parole e non parole), in which speed and accuracy scores were computed for pseudo-words reading (2 lists of 30 pseudo-words varying for length: short vs. long).

SECONDARY OUTCOMES:
Lexical access | 3 weeks
  Rapid automatized naming ability was assessed using the 'Rapid Automatized Naming test (RAN) - Colours' test (Test di denominazione rapida - Colori); in this test, matrices of 5 different colours were presented. The colours were presented in small 1 by 1 cm squares; they were black, blue (RGB 51-102-255), red (RGB 221-8-6), yellow (RGB 252-243-5), or green (RGB 31-183-20). There were 10 rows of 5 stimuli in each matrix for a total of 50 stimuli. Two different matrices for each condition were provided. In the RAN test, the child was requested to name each stimulus in the matrix as quickly and as accurately as possible. The dependent measure was the mean time in seconds/syllable. Naming errors were also recorded.
Phonological awareness: phonemic blending | 3 weeks
  Phoneme Blending assesses the capacity to derive a phonemic pattern from distinct phonemic units. The examiner presents each of 20 words, letter by letter, and the child is requested to mentally assemble them and report the resulting word. For both tasks, the scores refer to the total number of errors. Only age means (as raw scores) are provided.
Phonological awareness: phonemic elision | 3 weeks
  Phonemic Elision assesses the ability to recognize and isolate the phonemic constituents of 20 words (in this specific case, the initial constituents). The child is asked to delete the first two phonemes in the word read by the examiner and to report the resulting pseudo-word.
Auditory attention | 3 weeks
  Auditory selective attention was assessed using the Selective Auditory Attention Test from 'NEPSY-II'. In this task, the child listens to a pre-recorded list of words and touches the appropriate circle in the stimulus book when he or she hears a target word. This subtest has two parts. Auditory Attention is designed to assess selective auditory attention and the ability to sustain it (vigilance). Response Set is designed to assess the ability to shift and maintain a new and complex set involving both inhibition of previously learned responses and correctly responding to matching or contrasting stimuli. The child listens to a series of words and touches the appropriate circle when he or she hears a target word. Points are awarded only if the child responds correctly within 2 seconds of the target word presentation. Standard Scores are provided for the sum of Auditory Attention and Response Set.
Rhythm perception and reproduction | 3 weeks
  Rhythm and sound length discrimination abilities were assessed using the Rhythm Task from the 'Q1 VATA Assessment Battery for Cross-domain Learning Abilities' (Batteria per la valutazione delle abilità trasversali all'apprendimento, Q1 VATA). Subtest 'Duration' proposes sequences of tones for which the child has to identify and indicate the tone differing from the others in duration (being shorter or longer than the other tones). There are 4-5 tones in a sequence. In the 'Rhythm' subtest, the child listens to sequences of 6 to 10 tones that can be either identical or different in the rhythmic pattern, and he has to decide whether the two sequences are the same or different. Rhythm reproduction ability was measured using the 'Rhythm reproduction task' test (Tre prove di ritmo), which consists of the request to reproduce a set of rhythmic patterns of increasing complexity. The child has to reproduce a sequence of beats (with the top of a pencil) as demonstrated by the examiner.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Cancer, MD, Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Unit of Child Psychopathology, Scientific Institute IRCCS 'Eugenio Medea', Bosisio Parini, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cancer A, Bonacina S, Antonietti A, Salandi A, Molteni M, Lorusso ML. The Effectiveness of Interventions for Developmental Dyslexia: Rhythmic Reading Training Compared With Hemisphere-Specific Stimulation and Action Video Games. Front Psychol. 2020 Jun 3;11:1158. doi: 10.3389/fpsyg.2020.01158. eCollection 2020. PMID 32581961